CLINICAL TRIAL: NCT04151186
Title: A Clinical Study on the Safety and Efficacy of Chimeric Antigen Receptor T-cell Therapy for the TM4SF1- and EpCAM-positive Recurrent/Refractory Solid Tumors
Brief Title: A Clinical Study on the Safety and Efficacy of CAR-T Therapy for the TM4SF1- and EpCAM-positive Solid Tumors
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: suhaichuan (Other)
Collaborators: Shanghai Biomed-union Biotechnology Co., Ltd. (Unknown)
Responsible Party: Sponsor-Investigator, suhaichuan, professor, Tang-Du Hospital
Organization: Tang-Du Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CART-TM4SF1/CART-EpCAM-CAN-01
Record Dates: First submitted 2019-10-29; First posted 2019-11-05 (Actual); Last update posted 2019-11-05 (Actual); Status verified 2019-11

CONDITIONS: Advanced Solid Tumor; Neoplasms
Keywords: CAR-T cells; Immunologic Factors; TM4SF1;EpCAM
MeSH Terms: conditions — Neoplasms | interventions — TM4SF1 protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TM4SF1 and EpCAM positive CAR-T cells for solid tumors (Experimental): The present study is proposed to study advanced malignant solid tumors in adults, and the three escalating doses, namely, 2.0~2.5. 4.0~5.0 and 8.0~10.0 (×10 ^6/kg), will be given.
  Interventions: Biological: TM4SF1- and EpCAM-positive chimeric antigen receptor T-cell therapy

INTERVENTIONS:
Biological: TM4SF1- and EpCAM-positive chimeric antigen receptor T-cell therapy — Specification: 30 mL-100 mL, cell density of about (1-10) x10^6 cells/ml in each bag, number of T-cells about (1-10) x10^8 cells.) 300 ml for each infusion.
  Storage: The prepared CAR T-cells are cryopreserved in a preserving medium . This product is manufactured under the current good manufacture practices (cGMP) conditions, with restrictions on chemical components, free from animal- or human-derived components and confirming to the United States Pharmacopeia (USP)<71> and <85> regulations.
  Preservation: The frozen CAR T-cells are preserved in the liquid nitrogen transfer tank.
  Usage: The frozen CAR T-cells are preserved at low temperature and transferred to the bedside. The cells are thawed by 36 degrees centigrade to 38 degrees centigrade. water bath. The frozen cells are gently massaged until complete thawing. Then they are transfused back to the patients intravenously. The transfusion will be finished within 5-10 min.

SUMMARY:
* Transmembrane 4 L Six Family Member 1 (TM4SF1) and Epithelial cell adhesion molecule (EpCAM) are both highly expressed in many epithelial-derived solid tumors.
* The Chimeric Antigen Receptor T-cells (CAR-T) that target TM4SF1 or EpCAM have been generated respectively in our good manufacturing practices (GMP) facility and their anti-tumor effects have been demonstrated in multiple in vitro and in vivo studies.
* Clinical studies are proposed here to evaluate the anti-tumor activity of these cell therapy products for treatment of patients with TM4SF1 or EpCAM positive tumors. In this study, the safety, tolerance, and preliminary efficacy of CART-TM4SF1 and CART-EpCAM cells will be examined inpatients with refractory/recurrent advanced pancreatic cancer, colorectal cancer, gastric cancer or lung cancer. And 9 patients for each cancer will be evaluated.
* Clinical and immunological responses will be evaluated about 30 days and last up to 2 years after CAR-T cell infusion.

DETAILED DESCRIPTION:
Background:

* While great progress has been made in CAR T-cell therapy for the treatment of hematologic malignancies, its use in solid tumors is still at the exploratory stage.
* Transmembrane 4 L Six Family Member 1 (TM4SF1) protein mediates signal transduction events that play a role in the regulation of cell development, activation, growth and motility. It is a cell surface antigen and is highly expressed in different carcinomas. Epithelial cell adhesion molecule (EpCAM),is a transmembrane glycoprotein of 40 kilodaltons (kDa). EpCAM is highly expressed in many epithelial-derived tumors, such as colon, stomach, pancreas, lungs, ovaries and breasts. Recently, EpCAM has been identified as the surface marker of circulating tumor cells (CTCs) and cancer stem cells (CSCs).
* The investigators have developed novel TM4SF1-targeting CAR T-cells (CART-TM4SF1 cells) and EpCAM-targeting CAR T-cells (CART-EpCAM cells) for solid tumor treatment. These engineered T-cells can target and kill the TM4SF1- or EpCAM-positive tumor cells in vitro or in mice. Both of the CAR molecules contain a safety switch based on epidermal growth factor receptor (EGFR) to ensure the safety.
* The investigators propose to investigate the feasibility, safety, and efficacy of CART-TM4SF1 cells and CART-EpCAM cells for solid cancers in patients.

Objectives:

Primary objectives:

1. To determine the safety/tolerance dosages and adverse effects of CART-TM4SF1 cells or CART-EpCAM cells in the treatment of TM4SF1- or EpCAM-positive recurrent/refractory advanced solid tumors.
2. To preliminarily evaluate the efficacy of CART-TM4SF1 cells and CART-EpCAM cells in the treatment of TM4SF1- and EpCAM-positive recurrent/refractory advanced solid tumors.

Secondary objectives:

1. To determine the pharmacokinetic (PK)/pharmacodynamic (PD) characteristics of CART-TM4SF1 cells and CART-EpCAM cells in humans.
2. To evaluate the overall survival (OS) and tumor regression after treatment.
3. To assess the life quality of patients

Study population:

The study population includes 72 patients with refractory/recurrent advanced solid tumors positive for TM4SF1 or EpCAM expressions, each cancer including 9 patients . Among these patients with pancreatic cancer, colorectal cancer, gastric cancer or lung cancer, 9 subjects will receive 3 escalating doses (3 subjects in each dosage group)and safety and preliminary efficacy evaluation.

Design:

* This is a single-center open-label clinical study.
* Recruit patients with refractory/recurrent pancreatic cancer, colorectal cancer, gastric cancer or lung cancer, with written consent for this study. Perform biopsy to determine the expression of TM4SF1 or EpCAM of the tumor with immuno-histochemistry (IHC).
* Collect peripheral blood mononuclear cell (PBMC) from the patients, isolate and activate the T cells and transfect them with TM4SF1, or EpCAM targeting CAR, expand the transfected T cells as needed, assess the quality and antitumor activity of the CAR-T products in vitro and then transfer them back the patients via systemic or local injections, and follow up closely to collect related results as needed.
* Clinical and immunological responses will be evaluated closely in about 30 days and last up to 2 years after back-transfusion.

ELIGIBILITY:
Inclusion Criteria:

1. Aged≥18 years old and ≤75 years old when signing the informed consent; regardless of gender;
2. Body weight>40kg;
3. Pathologically confirmed as pancreatic cancer, colorectal cancer, gastric cancer or lung cancer;
4. Recurrent/refractory solid tumors unresponsive to the current standard treatment;
5. At least one measurable lesion according to the RECIST 1.1 criteria, that is, the long diameter of the non-lymph-node lesion≥10 mm, or the short diameter of the lymph node lesion ≥15 mm on CT or MRI cross-sectional imaging; the longest axis of the measurable lesion≥10 mm on CT scan (slice thickness≤5 mm in CT scan);
6. Acceptable hemopoietic ability: absolute neutrophil count (ANC) >1.5×10^9/L, platelet count >1.0×10^11/L, hemoglobin (HGB) >90g/L (no blood transfusion within two weeks), absolute lymphocyte count (ALC )>500×10^9/L;
7. Acceptable liver and kidney functions: aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5 ULN in subjects without liver metastases and ≤3.5 upper limit of normal (ULN) in those with liver metastases; bilirubin≤1.5 ULN (excluding hyperbilirubinemia or non-liver-derived hyperbilirubinemia); creatinine ≤1.5 ULN and creatinine clearance rate≥40 mL/min;
8. prothrombin time (PT)/international normalized ratio (INR) <1.5 ULN and partial thromboplastin time (PTT)/activated partial thromboplastin time (APTT) <1.5 ULN;
9. Positive for TM4SF1 or EpCAM expression (expression≥25%), with three classifications; (1) Recurrent or existing lesions at the primary site with tumor tissue samples collected within 1 year, which are positive for TM4SF1 or EpCAM by immunohistochemistry; (2) New metastatic lesions at the non-primary sites, which are positive for TM4SF1 or EpCAM by immunohistochemistry; (3) Remaining tumor lesions at the primary site with tumor tissue samples collected more than 1 year ago, and the lesions are positive for TM4SF1 or EpCAM by immunohistochemistry based on re-biopsy.
10. Women of child-bearing age (15-49 years old) must be negative for pregnancy test at 7 days before initiation of the treatment.
11. Eastern Cooperative Oncology Group (ECOG) scores≤2.
12. Expected survival no less than 12 weeks.

Exclusion Criteria:

1. History of any radiotherapy and chemotherapy within 4 weeks before a single blood collection;
2. History of any anti-programmed cell death protein 1 (PD1) and anti-Programmed cell death 1 ligand 1 (PD-L1) treatments within 12 weeks before a single blood collection;
3. History of organ transplantation;
4. Pregnancy or lactation;
5. Uncontrolled infectious diseases, such as baseline hepatitis B virus (HBV) DNA≥2000 IU/ml, positive for anti-human immunodeficiency virus （HIV） antibody and hepatitis C virus (HCV)-RNA;
6. Other active infection with clinical significance;
7. History of other active malignancies in the past 5 years, excluding basal or squamous skin carcinoma, superficial bladder cancer, and breast cancer in situ which have completely healed and require no follow-up treatment;
8. Serious autoimmune diseases or immunodeficiency disease, including those with confirmed severe autoimmune diseases and requiring long-term use (over 2 months) of systemic immunosuppressants (steroids) or having immune-mediated symptomatic diseases, such as ulcerative colitis, Crohn's disease, rheumatoid arthritis, systemic lupus erythematosus (SLE) and autoimmune vasculitis (eg., Wegener's granulomatosis);
9. Allergic diathesis and allergic to immunotherapy or relevant drugs;
10. Organ failure; Heart: Grade III and IV ; or with hypertension uncontrolled by the standard treatment, history of myocarditis or myocardial infarction within 1 year; Liver: Class C according to the Child-Turcottei-Pugh System (CTP); Kidneys: Kidney failure and uremic syndrome; Lungs: Serious symptoms of respiratory failure; Brain: Disturbance of consciousness;
11. Active bleeding, and thrombotic diseases requiring treatment;
12. Uncontrollable pleural and peritoneal effusion requiring clinical treatment or intervention;
13. T-cell cancers, such as T-cell lymphoma;
14. Current on systemic steroid or steroid inhalers;
15. Any mental diseases, including dementia and changes in mental status that may influence the understanding about the informed consent and questionnaire;
16. Participating in other clinical trials in the past 30 days;
17. Judged as serious uncontrollable diseases by the researchers, or other conditions that may interfere with the treatment and therefore being ineligible.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2019-11-20 (Estimated); Primary Completion 2021-05-20 (Estimated); Study Completion 2021-11-20 (Estimated)

PRIMARY OUTCOMES:
Safety assessed by Incidence of Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs) | 2 years
  1. After CAR-T cell infusion,the investigators will observe the potential adverse events related to the CAR-T cells infusion such as high fever, kidney failure and so on.
  2. Adverse events are coded according to MedDRA 22.0. List total number of AEs and SAEs; Number of subjects with different types of AEs and SAEs, case-times and incidence.AEs and SAEs are graded by National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTC AE version 5.0).

SECONDARY OUTCOMES:
CAR-T cell testing | 2 years
  The level of CAR-T cells will be tested regularly by Real-time Quantitative Polymerase Chain Reaction Detecting System(qPCR) or Flow cytometry to evaluate the proliferation in vivo and long-term survival
Overall response rate (ORR) | 2 years
  The ORR is defined as the percentage of participants who achieve partial response (PR) or better according to Response Evaluation Criteria In Solid Tumors（RECIST) criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Helong Zhang, professor, Study Chair — IEC of Institution for National Drug Clinical Trials ,Tangdu Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Visintin A, Knowlton K, Tyminski E, Lin CI, Zheng X, Marquette K, Jain S, Tchistiakova L, Li D, O'Donnell CJ, Maderna A, Cao X, Dunn R, Snyder WB, Abraham AK, Leal M, Shetty S, Barry A, Zawel L, Coyle AJ, Dvorak HF, Jaminet SC. Novel Anti-TM4SF1 Antibody-Drug Conjugates with Activity against Tumor Cells and Tumor Vasculature. Mol Cancer Ther. 2015 Aug;14(8):1868-76. doi: 10.1158/1535-7163.MCT-15-0188. Epub 2015 Jun 18. PMID 26089370
- [Background] Gao C, Yao H, Liu H, Feng Y, Yang Z. TM4SF1 is a potential target for anti-invasion and metastasis in ovarian cancer. BMC Cancer. 2019 Mar 15;19(1):237. doi: 10.1186/s12885-019-5417-7. PMID 30876464
- [Background] Peng XC, Zeng Z, Huang YN, Deng YC, Fu GH. Clinical significance of TM4SF1 as a tumor suppressor gene in gastric cancer. Cancer Med. 2018 Jun;7(6):2592-2600. doi: 10.1002/cam4.1494. Epub 2018 Apr 17. PMID 29665316
- [Background] Wang Y, Chen M, Wu Z, Tong C, Dai H, Guo Y, Liu Y, Huang J, Lv H, Luo C, Feng KC, Yang QM, Li XL, Han W. CD133-directed CAR T cells for advanced metastasis malignancies: A phase I trial. Oncoimmunology. 2018 May 7;7(7):e1440169. doi: 10.1080/2162402X.2018.1440169. eCollection 2018. PMID 29900044
- [Result] Hellstrom I, Horn D, Linsley P, Brown JP, Brankovan V, Hellstrom KE. Monoclonal mouse antibodies raised against human lung carcinoma. Cancer Res. 1986 Aug;46(8):3917-23. PMID 3731064
- [Result] Hellstrom I, Beaumier PL, Hellstrom KE. Antitumor effects of L6, an IgG2a antibody that reacts with most human carcinomas. Proc Natl Acad Sci U S A. 1986 Sep;83(18):7059-63. doi: 10.1073/pnas.83.18.7059. PMID 3462743
- [Result] Goodman GE, Hellstrom I, Brodzinsky L, Nicaise C, Kulander B, Hummel D, Hellstrom KE. Phase I trial of murine monoclonal antibody L6 in breast, colon, ovarian, and lung cancer. J Clin Oncol. 1990 Jun;8(6):1083-92. doi: 10.1200/JCO.1990.8.6.1083. PMID 2161448
- [Result] Goodman GE, Hellstrom I, Yelton DE, Murray JL, O'Hara S, Meaker E, Zeigler L, Palazollo P, Nicaise C, Usakewicz J, et al. Phase I trial of chimeric (human-mouse) monoclonal antibody L6 in patients with non-small-cell lung, colon, and breast cancer. Cancer Immunol Immunother. 1993;36(4):267-73. doi: 10.1007/BF01740909. PMID 8382560